CLINICAL TRIAL: NCT01002352
Title: Bariatric Outcomes Longitudinal Database (BOLD)
Acronym: BOLD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Surgical Review Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: BOLD
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Obesity; Overweight; Diabetes
Keywords: obesity; bariatric; BOLD; weightloss; database; data registry
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the Bariatric Outcomes Longitudinal Database (BOLD) study is to assess the mid- and long-term outcomes of bariatric surgeries and to analyze the relationship between these outcomes and 1) patient demographics and comorbidities, 2) clinical and surgical characteristics, and 3) pre-operative, peri-operative and post-operative care and treatment.

DETAILED DESCRIPTION:
Participants in the BOLD study include all patients who 1) have their bariatric surgery performed by either a Participant in the American Society for Metabolic and Bariatric Surgery designated Bariatric Surgery Center of Excellence or by a Fellow of the American Society for Metabolic and Bariatric Surgery 2) have been provided with a copy of the BOLD Patient Information Sheet. Patients under 18 years of age are included if a copy of the Patient Information Sheet is provided to an authorized legal representative.

The Patient Information Sheet containing information pertaining to the BOLD study is provided to the patient at the first pre-operative visit. The patient is not required to sign a consent form to participate in the study but must let the bariatric surgeon staff know if he/she does not wish to participate.

The following information will be collected for every bariatric surgery patient:

* Personal information: gender, race, employment status, insurance status, medical record number, year of birth, height, weight and prior surgeries. The surgeon has the option of entering patient name for internal tracking purposes.
* Information about surgery: date of admission, date of surgery and date of discharge.
* Information about medical condition before, during and after surgery.

Patient information is entered into BOLD through a secure website and permanently stored in a database that is managed by Surgical Review Corporation (SRC). This database is secure and meets the requirements for the protection of patient confidentiality as required by the Health Insurance Portability and Accountability Act (HIPAA).

Data that is used for research does not include the patient name or medical record number. Information about the patient's surgery will be combined with data from all other study participants in a separate research database and SRC research staff will analyze this combined information. The results of the study will be reported or published for the total population - no individual patient information will be published.

Surgeons participating in the study will attempt to obtain follow-up data on all patients who had surgery once a year for a minimum of at least five years following the date of surgery. Follow-up data can be obtained by the operating surgeon or designee, or by the patient's primary care physician and reported to the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery patients
* Males and Females
* All races

Exclusion Criteria:

* Negative psychological evaluation
* Surgeon's evaluation that patient is not a candidate for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who qualify for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2007-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of comorbidities | Within 1 year

SECONDARY OUTCOMES:
Mortality, weight loss, surgical complications | Within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Winegar, PH.D., Principal Investigator — Surgical Review Corporation
Locations (1):
- Surgical Review Corporation, Raleigh, North Carolina, United States

REFERENCES:
- [Derived] Li W, Gorecki P, Semaan E, Briggs W, Tortolani AJ, D'Ayala M. Concurrent prophylactic placement of inferior vena cava filter in gastric bypass and adjustable banding operations in the Bariatric Outcomes Longitudinal Database. J Vasc Surg. 2012 Jun;55(6):1690-5. doi: 10.1016/j.jvs.2011.12.056. Epub 2012 Feb 22. PMID 22360915
- See also: Surgical Review Corporation — http://www.surgicalreview.org